CLINICAL TRIAL: NCT03530137
Title: Collaboration to Promote Early Childhood Well Being in Families Experiencing Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00094422
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-06

CONDITIONS: Families Experiencing Homelessness With Children Under 48 Months of Age
Keywords: homelessness; homeless children; homeless families

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- families living at Families Moving Forward (FMF) (Other)
  Interventions: Behavioral: Healthy Home; Behavioral: Attachment and Biobehavioral Catch-up Infant (6-24 months) and Toddler (24-48 months).; Behavioral: HealthySteps

INTERVENTIONS:
Behavioral: Healthy Home — An evidence-based health literacy curriculum will be developed and implemented based on competencies of understanding and applying health information. The
Behavioral: Attachment and Biobehavioral Catch-up Infant (6-24 months) and Toddler (24-48 months). — ABC includes 10 in-home, manualized sessions with parents and infants, targeting: 1) increasing parents' nurturing when children are distressed, 2) helping parents follow children's lead, 3) decreasing frightening parent behaviors, and (for ABC-Toddler) managing dysregulation.
Behavioral: HealthySteps — Healthy Steps helps families identify, understand and manage parenting challenges like feeding, behavior, sleep, development and adjusting to life with a young child

SUMMARY:
The purpose of this study is to help us learn what are the best services to promote young children's healthy development for families who are experiencing homelessness. Participants may participate in three programs: 1. Healthy Home: four weekly, one-hour group sessions on health topics; 2. Attachment and Biobehavioral Catch-up (ABC): 10, one-hour parenting with parent and child; 3. Healthy Steps: helps families identify, understand and manage parenting challenges completed at well child visits. Participants will be asked to complete surveys, participate in focus groups, and interviews about the experiences with the services offered. Questionnaires about understanding health issues and surveys about parenting behaviors and self-efficacy will also be completed. Study duration is approximately 10 - 12 weeks. Programs may be continued once families move into permanent housing.

ELIGIBILITY:
Inclusion Criteria:

* Head of household of families living at FMF with at least one child under 48 months.
* All subjects must be English speaking and able to give legally effective consent.

Exclusion Criteria:

* Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured by a composite of satisfaction surveys and focus groups with families and staff. | up to 12 months
Changes in parent and child functioning as measured by composite of observation and self-report. | Baseline and 12 months

SECONDARY OUTCOMES:
Sustainability as measured by focus groups of staff | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Edie, DNP, Principal Investigator — Duke University; Karen A Carmody, PhD, Principal Investigator — Duke University
Locations (1):
- Families Moving Forward, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No